CLINICAL TRIAL: NCT01718132
Title: Reduction of Postoperative Pain, Nausea and Vomiting
Status: Completed | Type: Observational
Sponsor: Triemli Hospital (Other)
Responsible Party: Principal Investigator, Christoph K Hofer, Prof. Dr. med., Triemli Hospital
Other Study IDs: AWR-2012-STZ; KEK-StV-Nr. 47/12 (Other: ethic committee)
Record Dates: First submitted 2012-10-27; First posted 2012-10-31 (Estimated); Last update posted 2012-10-31 (Estimated); Status verified 2012-10

CONDITIONS: Post Operative Pain; Nausea and Vomiting
Keywords: Quality of the anaesthetic care in a PACU; reduction of postoperative pain; reduction of postoperative nausea and vomiting; quality markers
MeSH Terms: conditions — Pain, Postoperative; Nausea; Vomiting

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- postoperative patients

SUMMARY:
Aim of this prospective study was to assess the quality of postoperative care in a postoperative anaesthesia care unit (PACU) using postoperative pain, nausea and vomiting as well as their reduction as quality markers. So far, only sparse data related to this topic are available and there are currently no established quality markers of a PACU service.

ELIGIBILITY:
Inclusion Criteria:

All patients that have been transferred to the postanesthesia care unit postoperatively

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients that have been transferred to the postanesthesia care unit postoperatively
Sampling Method: Probability Sample
Enrollment: 16309 (Actual)
Dates: Start 2009-01; Primary Completion 2011-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Pain

SECONDARY OUTCOMES:
Postoperative nausea and vomiting

CONTACTS AND LOCATIONS:
Locations (1):
- Triemli City Hospital, Zurich, Switzerland